CLINICAL TRIAL: NCT00306579
Title: Myocardial Damage In Patients With Cerebral Infarction. Prevalence and Characteristics as Measured by Troponins, Electrocardiographic Changes and Myocardial Perfusion Imaging.
Brief Title: Myocardial Damage In Patients With Cerebral Infarction
Status: Completed | Type: Observational
Sponsor: Danish Heart Foundation (Other)
Collaborators: Fonden for Lægevidenskabelig Forskning for Fyns Amt. (Unknown); Novo Nordisk A/S (Industry); AJ Andersen og Hustrus Fond (Other); Overlægerådet Legatudvalg (Unknown); Raimond and Dagmar Ringgård-Bohn's Foundation (Other); Bankdirektør Hans Stener og hustru Agnes Steners legat (Unknown); Odense University Hospital (Other)
Other Study IDs: 054B26A43722225
Record Dates: First submitted 2006-03-23; First posted 2006-03-24 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; Myocardial ischemia; Myocardial necrosis
MeSH Terms: conditions — Ischemic Stroke; Myocardial Ischemia; Myocardial Infarction

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Introduction

For several years "ischemic" electrocardiographic (ECG) changes in the acute phase of ischemic stroke have been reported. Whether these ECG changes reflect true myocardial ischemia remains controversial. So far no study has assessed different markers of myocardial ischemia or necrosis in consecutive patients admitted to hospital with an acute ischemic stroke.

Purpose

The main purpose of this study is to determine the potential burden of reversible and irreversible myocardial ischemia in patients with an acute ischemic stroke.

Patients and methods

Serial blood samples for measuring troponin T, CK-MB and NT-proBNP are collected in 250 patients with evidence of an acute ischemic stroke admitted to the Department of Neurology at Odense University Hospital. In addition resting 12-lead ECG recordings will be obtained on a daily basis, and a 24-hour ST-segment ambulatory monitoring will be performed once within the first week of hospitalisation. Finally, myocardial perfusion patterns during rest will be evaluated by means of a myocardial perfusion scintigraphy in patients with an elevated troponin T level.

Six months later control measurements of troponin T, CK-MB and NT-proBNP and a 12-lead ECG will be obtained.

Expectations

The study will contribute with original observations in patients with acute ischemic stroke considering the following issues:

1. The prevalence and characteristics of ECG changes suggestive of myocardial ischemia.
2. The prevalence of transient ST-segment changes on ambulatory monitoring.
3. The prevalence and degree of myocardial necrosis as judged from biochemical markers.
4. The prevalence of reversible and irreversible perfusion defects on myocardial scintigraphy.
5. The prevalence, size and patterns of NT-proBNP.
6. Whether there is a change in ECG and biochemical markers over a 6-month follow-up period.

The results may have clinical implications regarding early and late treatment as well as clinical follow-up of patients recovering from an episode of acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke.
2. Age ≥ 18 years old.
3. Written, informed consent.

Exclusion Criteria:

1. Onset of stroke symptoms 8 to 21 days before admission.
2. Transient ischemic attack.
3. Intracerebral or subarachnoid haemorrhage.
4. Previous myocardial infarction.
5. Any pathological Q waves on the baseline ECG.
6. Current atrial fibrillation.
7. Unstable angina pectoris ≤ 3 weeks before admission.
8. Systolic blood pressure ≤ 90 mmHg and symptoms.
9. Resuscitation after cardiac arrest.
10. Unwillingness to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2003-08; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Jesper K. Jensen, MD, Principal Investigator — Department of Cardiology, Odense University Hospital; Hans Mickley, DMSci, Study Director — Department of Cardiology, Odense University Hospital; Søren Bak, MD, PhD, Study Chair — Department of Neurology, Odense University Hospital; Poul Flemming H. Carlsen, DMSci, Study Chair — Department of Nuclear Medicine, Odense University Hospital; Søren R. Kristensen, DMSci, Study Chair — Department of Clinical Chemistry, Aalborg Hospital